CLINICAL TRIAL: NCT05226910
Title: Transcranial Direct Current Combined With Intensive Therapies in Infantile Hemiplegia. Triple-blind Randomized Clinical Trial
Brief Title: HEMI-STIM. tDCS and Intensive Therapies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Rpalomo01
Record Dates: First submitted 2022-01-14; First posted 2022-02-07 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Infantile Hemiplegia
Keywords: infantile hemiplegia; upper extremity; transcranial direct current; children
MeSH Terms: conditions — Hemiplegia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Two groups: tDCS and Intensive therapies (experimental group), placebo and intensive therapies (control group)
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: It is a blind triple randomized clinical trial where patients, families and assessors are blinded and they do not know if the child is with placebo or current while is performing intensive therapies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS and intensive therapies (Experimental): Cathodal tDCS and constraint induce movement therapy
  Interventions: Device: tDCS and intensive therapies
- Sham and intensive therapies (Sham Comparator): Sham tDCS and constraint induce movement therapy
  Interventions: Device: Sham and intensive therapies

INTERVENTIONS:
Device: tDCS and intensive therapies — This intervention will consist in the combination of tDCS with CIMT (30 hours) and then with BIT (3 hours and 45 minutes)
  Arms: tDCS and intensive therapies
Device: Sham and intensive therapies — This intervention will consist in the combination of sham tDCS with CIMT (30 hours) and then with BIT (3 hours and 45 minutes)
  Arms: Sham and intensive therapies

SUMMARY:
Application of Transcranial Direct Current or placebo combined with Constraint Induced Movement Therapy (CIMT) and bimanual intensive therapy (BIT) in infantile hemiplegia (4-8 years). Before, after the treatment and 3 months after the treatment, the functionality of the affected upper limb will be assessed: Spontaneous use, alignment of the affected segment in movement, action of grasping and releasing an object with the wrist in a neutral position, extension and flexion and quality of life. CIMT will last 3 hours per day in a period of two weeks (10 days from M-F), and the transcranial direct current or placebo will be combined during the first 20 minutes of it. In addition, 45 minutes of BIT will be performed during the third week (3 days). The total time of the therapy will be 33 hours and 45 minutes. CIMT and BIT will have a playful and group performance model.

DETAILED DESCRIPTION:
Objectives: To determine the efficacy of the combined application of transcranial direct current (tDCS) with a restraint-induced movement therapy program and bimanual therapy on quality of life, quality of movement and spontaneous use of the affected upper limb in children. with infantile hemiparesis.

Design: Randomized clinical trial with triple blind placebo control. Participants: 30 children between 4 and 8 years old diagnosed with infantile hemiparesis randomized into two groups.

Intervention: Program of 15 sessions (3 weeks) in which 20 minutes of cathodic tDCS (active or placebo) will be applied during the performance of 3 hours of restriction-induced movement therapy (CIMT) in the first two weeks and with 45 minutes of bimanual intensive therapy (TIB) in the third week. The effective duration of the intervention will be 33 hours and 45 minutes.

Variables: The outcome variables will be recorded before the intervention program, just after and three months after its completion.

Analysis: An intention-to-treat analysis will be performed. For the main result variables, a two-factor ANOVA (intervention-time) will be performed with a post-hoc analysis with Bonferroni correction.

ELIGIBILITY:
Inclusion Criteria:

* Children between 4 and 8 years old, with a diagnosis of congenital infantile hemiplegia, with a score between levels I and III of the manual ability classification system (MACS) and a level I-III of the gross motor function classification system will be included (GMFCS). In addition, children must have a preserved cognitive ability to understand the execution of structured activities

Exclusion Criteria:

* Having previously been treated with tDCS; Having been infiltrated with botulinum toxin 2 months prior to the intervention; Surgery of the upper limb the 6 months prior to the intervention; Pharmacologically uncontrolled epilepsy or having suffered epileptic seizures in the two years prior to the study (according to international recommendations for tDCS in children, Gillick et al., 2018); Contraindications of tDCS according to international recommendations. In addition, a withdrawal criterion will be non-attendance for more than 20% of the hours of the program.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Change of the spontaneous use of affected upper limb | Baseline, post-treatment (at 13 days), and follow-up at 12 weeks
  This outcome will be assessed with Shuee evaluation. This evaluation uses the modified House scale which a maximum of 45 points can be obtained for the spontaneous use, and the values obtained can be converted into percentages. In addition, the dynamic positioning of the affected upper extremity is assessed through 16 structured activities in the Shuee evaluation (Positioning of the thumb, fingers, wrist, elbow, and forearm).
  TAcquiring a maximum score of 72 and their values can be considered in percentages. Another of the measured variables into the Shuee evaluation is the action of grasping and releasing an object with the wrist joint in different positions (results provided in percentages). This evaluation is validated for children with hemiplegia from 3 to 18 years old.

SECONDARY OUTCOMES:
Change in the experience of use of the affected upper limb | Baseline, post-treatment (at 13 days), and follow-up at 12 weeks
  This outcome will be assessed with CHEQ questionnaire. It is validated for children with have reduction in the upper limb from 8 to 18 years old. It is a questionnaire composed of 27 questions about the activities of daily life and the execution of the task. Whether it is done with one hand, with both hands or with help and how effective is the use of the affected hand on a scale of 1-4, the time of execution of the task on a scale of 1-4 and the discomfort of execution of it on a scale of 1-4. It can be answered by the family, the therapist or the child himself from the age of 13.
Change in the Quality of life in cerebral palsy | Baseline, post-treatment (at 13 days), and follow-up at 12 weeks
  Use the PedsQL questionnaire to measure the quality of life. It is a questionnaire answered by the parents with children with cerebral palsy from 2-18 years old. It is made up of 35 items that describe different situations in the child's life. The questionnaire has different domains related to the physical activities, school activities, emotional activities, hygiene. The maximum score obtained can be 100 (0-100), which indicates that the higher the score, the better the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Gómez-Soriano, PhD, Principal Investigator — Castilla-La Mancha University
Locations (1):
- University of Castilla-La Mancha, Toledo, Spain

IPD SHARING:
Plan to Share IPD: Yes
We will share all data researchers need
Supporting Information: ICF
Time Frame: Following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent ethical committee identified for this purpose.
  The proposal should be directed to principal investigator.

REFERENCES:
- [Background] Alisar DC, Ozen S, Sozay S. Effects of Bihemispheric Transcranial Direct Current Stimulation on Upper Extremity Function in Stroke Patients: A randomized Double-Blind Sham-Controlled Study. J Stroke Cerebrovasc Dis. 2020 Jan;29(1):104454. doi: 10.1016/j.jstrokecerebrovasdis.2019.104454. Epub 2019 Nov 4. PMID 31699572
- [Background] Page SJ, Cunningham DA, Plow E, Blazak B. It takes two: noninvasive brain stimulation combined with neurorehabilitation. Arch Phys Med Rehabil. 2015 Apr;96(4 Suppl):S89-93. doi: 10.1016/j.apmr.2014.09.019. PMID 25813373
- [Background] Hoare BJ, Wallen MA, Thorley MN, Jackman ML, Carey LM, Imms C. Constraint-induced movement therapy in children with unilateral cerebral palsy. Cochrane Database Syst Rev. 2019 Apr 1;4(4):CD004149. doi: 10.1002/14651858.CD004149.pub3. PMID 30932166
- [Background] Gordon AM, Hung YC, Brandao M, Ferre CL, Kuo HC, Friel K, Petra E, Chinnan A, Charles JR. Bimanual training and constraint-induced movement therapy in children with hemiplegic cerebral palsy: a randomized trial. Neurorehabil Neural Repair. 2011 Oct;25(8):692-702. doi: 10.1177/1545968311402508. Epub 2011 Jun 23. PMID 21700924